CLINICAL TRIAL: NCT04173403
Title: A Long-term Study to Evaluate the Efficacy and Safety of AK102 in Combination With Lipid-lowering Therapy in Patients With Hypercholesterolemia
Brief Title: A Long-term Study of AK102 in Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: AD Pharma (Guangdong) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK102-204
Record Dates: First submitted 2019-11-17; First posted 2019-11-22 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK102 (Experimental): 450mg AK102, Q4W, subcutaneous injection; OR 300mg AK102, Q4W, subcutaneous injection;OR 150mg AK102, Q4W, subcutaneous injection;
  Interventions: Drug: 450mg AK102; Drug: 300mg AK102; Drug: 150mg AK102; Drug: Statins and/or Ezetimibe

INTERVENTIONS:
Drug: 450mg AK102 — AK102 Q4W
Drug: 300mg AK102 — AK102 Q4W
Drug: 150mg AK102 — AK102 Q2W
Drug: Statins and/or Ezetimibe — Lipid-lowering therapies

SUMMARY:
This is a phase II, open-label, non-controlled, extended study. The main objective of this study is to evaluate the long-term efficacy and safety of AK102 in combination with basic lipid-lowering therapy in patients with hypercholesterolemia. Subjects who have participated in the AK102 studies and have completed the last visit,and who, in the opinion of the investigator, are likely to benefit from continued treatment will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Body weight ≥ 40 kg for both men and women.
3. Participated in the AK102-202 study, and completed the AK102-202 study last visit.

Exclusion Criteria:

1. Poor compliance in AK102-202 study per investigator's judgement.
2. AE that led to permanent discontinuation of AK102 occurred during the AK102-202 study period.
3. Prior use of PCSK9 inhibitors other than AK102.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 796 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 52 | Week 52

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events as assessed by CTCAE V5.0 | From baseline through 52 weeks
Percent Change From Baseline in High-density lipoprotein (HDL) cholesterol | From baseline through 52 weeks
Percent Change From Baseline in non High-density lipoprotein (non-HDL) cholesterol | From baseline through 52 weeks
Percent Change From Baseline in Serum Triglyceride (TG) cholesterol | From baseline through 52 weeks
Percent Change From Baseline in Apolipoprotein B (Apo B) | From baseline through 52 weeks
Percent Change From Baseline in Apolipoprotein A-I (Apo A-I) | From baseline through 52 weeks
Percent Change From BaPercent Change From Baseline in Total Cholesterol(TC) | From baseline through 52 weeks
Change From Baseline in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) | From baseline through 52 weeks
Concentrations of AK102 in Serum | From baseline through 52 weeks
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From baseline through 52 weeks
  The immunogenicity of AK102 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Shuyang Zhang, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No